CLINICAL TRIAL: NCT05491837
Title: Effects of Device Induced Acute Intermittent Hypoxia in Upper and Lower Limb Activity Functions in Persons With Incomplete Spinal Cord Injury.
Brief Title: Effects of Intermittent Hypoxia in Upper and Lower Limb Functions in Persons With Incomplete Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIPHAH/RCRS/REC/Letter-0129
Record Dates: First submitted 2022-07-24; First posted 2022-08-08 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Incomplete Spinal Cord Injury
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: The participants are randomly divided into 2 groups. Interventional and SHAM
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients 'selection and their allocation of treatments to experimental and control will be done by team of physiotherapists working in paraplegic center Peshawar who will not the part of investigation team. Treatment will be given by trained physiotherapist within paraplegic center Peshawar while data will be analyzed by statistician working in Riphah International University. The investigator, patients and the treatment providers will be anonymous from the group allocation, treatment they receive and data analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Interventional group will be provided a brief sequence of acute hypoxia consisting of 9% oxygen via device HYP 123 for one minute followed by normoxia 21% of oxygen for a total of 15 repetition.
  This protocols will be provided 3 times/week for a period of 4 weeks.
  Interventions: Other: Device induce acute intermittent hypoxia 9 % of Oxygen; Other: Normoxia 21% of oxygen
- Control group (Sham Comparator): SHAM group' participants will be provided 21% of O2 (normoxia), comprised of 15 repetitions of 1-minute then switching to another 1-minute of 21% O2.
  This protocols will be provided 3 times/week for a period of 4 weeks.
  Interventions: Other: Normoxia 21% of oxygen

INTERVENTIONS:
Other: Device induce acute intermittent hypoxia 9 % of Oxygen — Interventional group will be provided a brief sequence of mild hypoxia consisting of 9% oxygen for one minute followed by normoxia 21% of oxygen for a total of 15 episodes
  Arms: Interventional group
Other: Normoxia 21% of oxygen — SHAM group will be provided normoxia 21% of Oxygen

SUMMARY:
Spinal cord injury (SCI) is a devastating disability with physical, social and vocational consequences. Owing to its overwhelming complications, the cost of treatment and rehabilitation increases constantly. Persons with spinal cord injury are always dependent on their families in most of house hold, recreational and activities of daily life. Majority of SCI are incomplete classification C or D as per American spinal injury Association (ASIA). Due to certain spared pathways intrinsic mechanism of neuroplasticity take place in incomplete spinal cord injuries (iSCI) which is liable for natural recovery, but this potential is limited and often slow. Therefore there is need for some advance therapeutic interventions which may enhance neuroplasticity and improve functional recovery in individuals with iSCI.

It has been reported that acute intermittent hypoxia (AIH) increase neuro plasticity by causing release of spinal serotonin which stimulate serotonin type 2 (5-HT2) receptors that undergoes a series of mechanisms which increase brain derived neurotrophic factors (BDNF) which subsequently enhance motor functions of upper and lower limbs in iSCI.

Despite of the growing body of literatures supporting that AIH improves both upper limb and lower limb functions along with walking ability and speed. However, their results are limited to small sample size, gender biased and lack of intralimbs assessment. As per the author knowledge, these literatures lack retention effects of AIH on upper and lower limb function. In addition variables like quality of life, disability and some biomarkers related to hypoxic effects have not been reported in any of these studies. Furthermore, it is hypothesized that variant geographic locations and socioeconomic status may affects persons with iSCI differently. So in light of these literature gaps, the author aim is to investigate the effects of AIH in upper and lower limb motor function, balance, quality of life and disability. In addition, the effects of AIH on brain derived neurotrophic factors (BDNF), hemoglobin (Hb) level, numbers of RBS and hematocrits will be assessed.

DETAILED DESCRIPTION:
Study design and setting: This will be Randomized Controlled Trail triple blind study design. The study will be conducted in Paraplegic center Peshawar (PCP) Pakistan https://paraplegiccenter.org/.

Blinding of the participants: Patients 'selection and their allocation of treatments to experimental and control will be done by team of physiotherapists working in paraplegic center Peshawar whose will not the part of investigation team. Treatment will be given by trained physiotherapist within paraplegic center Peshawar while data will be analyzed by statistician working in Riphah international University Islamabad Pakistan. The investigators, patients and the treatment providers will be anonymous from the group allocation, treatment they receive and data analysis.

Sampling Technique: Since the sample frame is available so sample technique will be Random Sampling by computer generated table of random number.

Sample size: Sample size for the study calculated via G Power sample size calculator with power of 95% and α error probability is 0.05 on the following assumption.

Walking speed (10MWT) post intervention in groups are: IH= 17.1±5.8 vs. Nx=7.1±2.8s. the effect was determined as 2.09. So the total sample size for both groups is 8 (4). Since this sample size is less so we consider our effect size 0.9 thus total sample size will be 68, each grip will be having 34 participants.

Participants: Person with incomplete spinal cord injury will be our study participants.

Tools/Outcome measures include the following

1. Hypoxico Hyp 123
2. Hand Dynamometer (Grip strength) Hydraulic guage (pinch strength)
3. Upper limb functional Test (9-Hole and Pegs Test, Box and Block Test)
4. Quick-DASH (Disability of arm, shoulder and hand)
5. Ten Minute Walk Test ,Time up and Go Test (walking performance)
6. Six Minute Walk Test(endurance)
7. Berg Balance Test (Balance)
8. WHO-QOL (BREF Urdu version)
9. Brain derived neurotrophic factors (BDNF)
10. Level of Hemoglobin, RBS and Hematocrits Interventions details: After randomly allocation of the patients into intervention and SHAM group. The Interventional group will be provided a brief sequence of mild hypoxia consisting of 9% oxygen for one minute followed by normoxia 21% of oxygen for a total of 15 episodes. The SHAM group' participants will be provided 21% of O2 (normoxia), comprised of 15 repetitions of 1-minute then switching to another 1-minute of 21% O2. Both these protocols will be provided 3 times/week for a period of 4 weeks. Both groups will continue their routine rehabilitation for the upper and lower limb exerccises within the center. Post assessments for the said variable will be carried out each week (post 7 days, post 14 days, post 21 days, post 30 days and a follow up week for retention effects).

Data collection Procedure: After informed consent, all the willing and eligible participants will be randomly divided into intervention and SHAM group. Participant's demographic details will be taken which includes participant's age, geographic location, socioeconomic status, history of onset of iSCI, level of spinal cord injury, ASIA classification C/D and BMI. Outcome measure will be assessed as baseline at each week and after final as retention effect ass discussed above.

Ethical consideration: Ethical consideration has been provided by the ethical board of Riphah International University Islamabad RIPHAH/RCRS/REC/Letter-0129 dated march 2022.

ELIGIBILITY:
Inclusion Criteria:

1. Incomplete SCI≥ 3 months(21);
2. Traumatic and non-traumatic, non-progressive lesions, Aged ≥ 18 years ;
3. LesionC4 and below as classified ASIA category C and D;
4. Both gender
5. Ability to ambulate with or without assistive devices; and
6. Ability to follow verbal and visual command.

Exclusion Criteria:

1. Participants with complete spinal cord injury;
2. Unstable orthopedic injuries and joint contractures
3. Osteoporosis with high risk of fracture;
4. Pressure ulcers and cutaneous lesion(4)
5. Cognitive impairment, severe cardiopulmonary complication such as severe breathing disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-04 (Estimated)

PRIMARY OUTCOMES:
Upper limb function | change will be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  Change in upper limb function will be assessed via 9-Hole peg test (9-HPT) and Box and Block test (BBT).The 9-HPT is used to assess fine movement of hand and finger dexterity. It has excellent reliability and adequate to good concurrent validity with Box and Block test. It should be conducted with the dominant hand first. The participants will be advised to place the pegs into the 9 hole in the board and then again remove each peg and place it in the container. Total time will be measured and it will be compared with the other hand. The BBT is used to test manual dexterity. The participants are requested to move 1 inch block from one box to another in 60 seconds while crossing the partition between the blocks. Total blocks moved will be calculated as test score.
upper limb grip strength | change in grip strength will be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  change in Grip strength will be measured by using hand dynamometer (Model-Jamardigital Hand dynamometer). Participants will be seated with shoulder adducted and neutral rotated, elbow at 90 degree position. The forearm is in between supination and pronation without support of arm rest and the wrist is in neutral position. Maximum contraction will be measured by asking the participants to contract against the hand grip while maintaining the contraction for 3 to 5 seconds. Average of 3 attempts will be calculated as measurement
Upper limb Pinch strength | change in pinch strength will be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  change in Pinch strength will be measured by using hydraulic gauge. Hydraulic gauge for pinch strength is reliable with ICC 0.821. Pinch strength is used incomplete spinal cord injury tetraplegic populations. The patient is advised to apply force on pinch grove within the device and then gauge will calibrate the total force in pounds or kilograms. All type of pinch strength will be measured and score will be compared with the normal values.
Quick DASH to measure upper limb disability | It will be assed on baseline and after 4 week of interventions
  Quick Disability of arm, shoulder and Hand (DASH) questionnaire is a self-reporting 11-items questionnaire that measures the ability of patients to perform certain upper limb tasks. The patients can rate their difficulty that they may face during specific upper limb activity on 5 points likert scale. The questionnaire is designed to assess one or more disability of arm shoulder and hand. It has good validity and reliability. The interclass correlation coefficient (ICC) is 0.82 The test retest reliability of the both 11 item and its optional work 15 items are 0.9 and 0.94 respectively and that neither of them are significant difference from that of the original DASH questionnaire
walking performance | change in walking performance will be measured on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  Change in walking performance will be assessed via 10 meter 'walk test(10MWT). It is used to assess walking performance of individual. It measures times in seconds the participants is taken during 10 meters of walking as quickly as possible using their regular devices. This scale has been validated for iSCI and its test retest, intra-rater are excellent (r= 0.983) while inter-rater r=0.97.
  The Time up and go test (TUG)is used to evaluate the walking performance of an individual that he takes to stand up from chair and walk 3 meters independently with her/his own pace of walking. Then return to resume his seated position again. Total time in seconds will be calculated. This scale has excellent validity and both test retest and intra rater reliability r=0.98 while inter-rater reliability reported as r=0.97.
walking endurance | change will be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  Chane in walking endurance will be measured via 6 minute walk test. This scale is validated for patients with iSCI with an excellent inter rater reliability r- 0.98. The participants are advised to walk 6 minutes as far as possible in 6 minutes while total distance in meters is calculated. Participants can rest if needed but they are advised not to sit
lower limb muscle strength | change in lower limb strength be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  Lower limb dynamometer is used to quantify strength of lower limb muscles. It assesses isometric strength of lower limb muscles and considered a suitable alternative of conventional manual muscle testing.
balance | change in balance score will be assessed on base line before intervention, post 7 days, post 14 days, post 21 days, post 30 days and a follow up week without intervention for retention effects
  The berg balance scale(BBS) was originally developed for stroke and geriatric population but it's used is also evident in iSCI(40). It is 14-items scale that is used to assess static balance and fall risk in adults. It has been used in various neurological disorders. In incomplete spinal cord injury, it is reported that BBS has excellent inter-observer reliability both for single item and for total items r =.84 and ICC =0.95 (41). The concurrent validated of BBS in regard to spinal cord injury is also reported moderate to high (40). The BBS total score is 56 and less than 45 indicated risk of fall
Brain derived Neurotrophic factors (BDNF) to measure plasticity in brain | It will be assed on baseline and after 4 week of interventions
  Brain derived neurotrophic factors are secreted by the neuron which is one of the important factors in neural plasticity. Effects of various locomotor exercise in incomplete spinal cord injury have been investigated. It is premised that BDNF activate high affinity tropomyosin related kinase receptor subtype B (TrKB) also called tyorosin kinase B that help in rhythmic activity of diagram in cervical incomplete spinal cord injury. In human, BDNFis present in blood platelets where it starts accumulating during synthesis of megakaryocytes. It can be readily detectable in human serum by ELIZA using monoclonal antibodies and thus it is considered reliable and has been largely speculated that it may improve brain functions

SECONDARY OUTCOMES:
WHO QOL Urdu version to assess quality of life | It will be assed on baseline and after 4 week of interventions
  WHOQOL-BREF is a short version of WHOQOL-100. It is widely used quality of life questionnaire in various conditions and applicable cross culturally. It comprises of four domains each incorporated with various facets to form 26 questions in total. It has been shown that its internal consistency is good Cronbach α range 0.74-o.78 in spinal cord injury

CONTACTS AND LOCATIONS:
Overall Officials: Ikram Ali, Master, Principal Investigator — Riphah International University Islamabad; Waqar Ahmed Awan, PhD, Study Chair — Riphah International University Islamabad
Locations (1):
- Riphah International University Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
At this stage IPD is No. Once the data collection process is started and individual consent form including their permission for publication of the data is taken. Then IPD will be shared accordingly.

REFERENCES:
- [Background] Ahuja CS, Wilson JR, Nori S, Kotter MRN, Druschel C, Curt A, Fehlings MG. Traumatic spinal cord injury. Nat Rev Dis Primers. 2017 Apr 27;3:17018. doi: 10.1038/nrdp.2017.18. PMID 28447605
- [Background] Yang R, Guo L, Wang P, Huang L, Tang Y, Wang W, Chen K, Ye J, Lu C, Wu Y, Shen H. Epidemiology of spinal cord injuries and risk factors for complete injuries in Guangdong, China: a retrospective study. PLoS One. 2014 Jan 28;9(1):e84733. doi: 10.1371/journal.pone.0084733. eCollection 2014. PMID 24489652
- [Background] Navarrete-Opazo A, Alcayaga J, Sepulveda O, Rojas E, Astudillo C. Repetitive Intermittent Hypoxia and Locomotor Training Enhances Walking Function in Incomplete Spinal Cord Injury Subjects: A Randomized, Triple-Blind, Placebo-Controlled Clinical Trial. J Neurotrauma. 2017 May 1;34(9):1803-1812. doi: 10.1089/neu.2016.4478. Epub 2016 Jul 19. PMID 27329506
- [Background] Champod AS, Eskes GA, Foster GE, Hanly PJ, Pialoux V, Beaudin AE, Poulin MJ. Effects of acute intermittent hypoxia on working memory in young healthy adults. Am J Respir Crit Care Med. 2013 May 15;187(10):1148-50. doi: 10.1164/rccm.201209-1742LE. No abstract available. PMID 23675727
- [Background] Manukhina EB, Downey HF, Shi X, Mallet RT. Intermittent hypoxia training protects cerebrovascular function in Alzheimer's disease. Exp Biol Med (Maywood). 2016 Jun;241(12):1351-63. doi: 10.1177/1535370216649060. Epub 2016 May 10. PMID 27190276
- [Background] Viscor G, Torrella JR, Corral L, Ricart A, Javierre C, Pages T, Ventura JL. Physiological and Biological Responses to Short-Term Intermittent Hypobaric Hypoxia Exposure: From Sports and Mountain Medicine to New Biomedical Applications. Front Physiol. 2018 Jul 9;9:814. doi: 10.3389/fphys.2018.00814. eCollection 2018. PMID 30038574
- [Background] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- [Background] Sandhu MS, Perez MA, Oudega M, Mitchell GS, Rymer WZ. Efficacy and time course of acute intermittent hypoxia effects in the upper extremities of people with cervical spinal cord injury. Exp Neurol. 2021 Aug;342:113722. doi: 10.1016/j.expneurol.2021.113722. Epub 2021 Apr 28. PMID 33932397
- [Background] Trumbower RD, Jayaraman A, Mitchell GS, Rymer WZ. Exposure to acute intermittent hypoxia augments somatic motor function in humans with incomplete spinal cord injury. Neurorehabil Neural Repair. 2012 Feb;26(2):163-72. doi: 10.1177/1545968311412055. Epub 2011 Aug 5. PMID 21821826